CLINICAL TRIAL: NCT06645132
Title: Pilot Study to Understand the Feasibility of Implementing a Wearable Device Cueing System Following Bone Marrow Transplant
Brief Title: Understanding the Implementation of Cued Exercise Using Wearable Devices and a Custom Smartphone Application Following Bone Marrow Transplant.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Whitney Morelli, Principal Investigator, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00051086
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-11

CONDITIONS: Blood Cancer; Bone Marrow Transplant (BMT)
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reminders to exercise through cues provided by wearable device + custom smartphone application (Experimental): Each participant receives 2 wearable devices and custom smartphone application. Participants will wear an activity monitor on their non-dominant wrist and contralateral ankle. Post-transplant inpatient days ~3-10, participants will schedule three cued exercise sessions each day using the smartphone application. At the scheduled time, the wearable devices will vibrate to indicate "time to exercise" and participants are encouraged to complete an exercise task for 15 minutes. Post-transplant inpatient hospital days ~1-2 and post-transplant inpatient hospital days ~11 until discharge patients will wear the devices but will not receive any cues. During these days, the monitors will only be measuring their movement without any intervention.
  Interventions: Behavioral: exercise intervention

INTERVENTIONS:
Behavioral: exercise intervention — Exercise intervention leveraging wearable devices and a custom smartphone application to cue exercise as a reminder during idle time during an inpatient hospital stay, post allogenic bone marrow transplant.

SUMMARY:
The purpose of this study is to pilot test the feasibility of providing patients diagnosed with a hematologic malignancy, undergoing an allogeneic bone marrow transplant, a wearable device and smartphone app (similar to a Fitbit), that would send personalized reminders to move during their post-transplant inpatient hospital stay to promote physical recovery and well-being.

DETAILED DESCRIPTION:
Enrolled patients who have been diagnosed with a hematologic malignancy and are scheduled to undergo an allogeneic bone marrow transplant will use a custom-designed wearable device and smartphone application as a behavioral intervention to cue exercise. Participants will be asked to wear the wearable device for the duration of their post-transplant inpatient hospital stay.

Aim 1. To examine the potential efficacy of the wearable device + smartphone application to prompt alloBMT patients to move.

Aim 2. To receive participant feedback on their experience participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosed with hematologic malignancy
* Scheduled to receive an alloBMT
* Physician consent to participate in the study

Exclusion Criteria:

• Inability to complete 15 minutes walking unassisted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pilot evaluation of intervention efficacy | cumulative percent from day 1 through discharge from hospital, on average day 30
  Efficacy will be evaluated by examining the percentage of time participants responded to the cued exercise prompts.
Patient feedback from participation in the study | day 10
  Patient experience will be evaluated by looking at the central tendencies of the ratings from the post-participation evaluation survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No